CLINICAL TRIAL: NCT07085117
Title: Real World Use, Effectiveness and Safety of Teprotumumab Among Thyroid Eye Disease Patients Treated in China BOAO Pilot Zone: A Retrospective Cohort Study
Brief Title: Real World Study to Describe the Effectiveness and Safety of Teprotumumab Among Thyroid Eye Disease Patients
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20240345; EUPAS1000000625 (Other: EU PAS number)
Record Dates: First submitted 2025-06-30; First posted 2025-07-25 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Thyroid Eye Disease
Keywords: Thyroid Eye Disease; Teprotumumab; TEPEZZA®
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — teprotumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Teprotumumab: Participants with Thyroid Eye Disease (TED) that have received teprotumumab treatment in BOAO Pilot Zone.
  Interventions: Drug: Teprotumumab

INTERVENTIONS:
Drug: Teprotumumab — Participants received teprotumumab as an intravenous (IV) infusion.
  Other Names: TEPEZZA®

SUMMARY:
The main objective of this study is to assess the number of participants with proptosis response as of last intravenous infusion of teprotumumab.

DETAILED DESCRIPTION:
A retrospective cohort will be followed retrospectively for endpoints at the only facility providing treatment of teprotumumab in mainland China. Eligible participants' data were collected retrospectively over a period of approximately 3 years. The target population is patients with Thyroid Eye Disease (TED) that have received teprotumumab treatment in BOAO Pilot Zone. While the primary objective is to assess the proportion of patients with proptosis response as of the last intravenous infusion of teprotumumab, the secondary objectives are to describe baseline characteristics of patients at teprotumumab initiation, and the teprotumumab use at follow-up, to describe real-world effectiveness of clinical outcomes of interest, to describe patient-reported outcomes and to describe real-world safety of teprotumumab.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of at least 1 infusion of teprotumumab for treatment of the TED.
* Obtained study specific informed consent form (ICF), if required.

Exclusion Criteria:

* Documentation of non-Chinese ethnicity.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with TED that have received teprotumumab treatment in BOAO Pilot Zone.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2025-07-02 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Proptosis Response as of the Last IV Infusion Teprotumumab | From baseline up to approximately 3 years
  Proptosis response is defined as having a ≥ 2 mm reduction in proptosis measurement from baseline in the more severely affected eye without deterioration (≥ 2 mm increase) of proptosis in the fellow eye following the last infusion.

SECONDARY OUTCOMES:
Demographics of Participants at Teprotumumab Initiation | From baseline up to approximately 3 years
  Demographics include age in years and sex (male, female, unknown).
Clinical Characteristics of Participants at Teprotumumab Initiation: Body Mass Index at Index Date | From baseline up to approximately 3 years
Clinical Characteristics of Participants at Teprotumumab Initiation: Smoking Status | From baseline up to approximately 3 years
Clinical Characteristics of Participants at Teprotumumab Initiation: Disease Duration | From baseline up to approximately 3 years
Clinical Characteristics of Participants at Teprotumumab Initiation: TED Activity | From baseline up to approximately 3 years
Clinical Characteristics of Participants at Teprotumumab Initiation: TED Severity | From baseline up to approximately 3 years
Clinical Characteristics of Participants at Teprotumumab Initiation: Eye symptoms | From baseline up to approximately 3 years
Clinical Characteristics of Participants at Teprotumumab Initiation: Clinical Activity Score | From baseline up to approximately 3 years
Clinical Characteristics of Participants at Teprotumumab Initiation: Computed Tomography (CT)/Magnetic Resonance Imaging (MRI) Measurements | From baseline up to approximately 3 years
Clinical Characteristics of Participants at Teprotumumab Initiation: Quality of Life | From baseline up to approximately 3 years
Number of Participants with Relevant Medical History at Teprotumumab Initiation | From baseline up to approximately 3 years
  Medical history includes history of compressive optic neuropathy, hyperglycemia, inflammatory bowel disease (IBD), infusion reactions, and hearing impairment; therapeutic history for thyroid disease (Graves' disease or others) before teprotumumab administration; therapeutic history for TED before teprotumumab administration and complications if any; comorbidities; concomitant treatments; lab tests.
Teprotumumab Use | From baseline up to approximately 3 years
  Teprotumumab use includes dose and dosing schedule, total number of infusions and duration, dose reduction and modification (including causes), treatment interruption and causes, time interval from interruption to re-initiation, and subsequent re-initiation treatment (if any), treatment discontinuation (including causes).
Proptosis Measurements of Participants | From baseline up to approximately 3 years
  Proptosis measurements include all available proptosis measurements by eye for each participant and the change in proptosis measurement between baseline and the last infusion by eye.
Clinical Activity Scores (CAS) of Participants | From baseline up to approximately 3 years
  CAS will include all available measures of CAS items by eye for each participant and the number of participants achieving CAS value of 0 or 1 as of the last infusion among patients with active TED at baseline.
Overall Response as of the Last Infusion Among Participants with Active TED | From baseline up to approximately 3 years
  Overall response is defined as having ≥ 2-point reduction in CAS AND ≥ 2 mm reduction in proptosis from baseline in the most severely affected eye, provided there is no corresponding deterioration (≥ 2-point increase in CAS or ≥ 2 mm increase in proptosis) in the fellow eye following the last infusion.
  Active TED is defined as CAS≥3 on a 7-point scale at baseline.
Diplopia Measurements for Participants | From baseline up to approximately 3 years
  Diplopia measurements will include all available measures of diplopia for each participant, the binocular diplopia response as of the last infusion defined as having baseline binocular diplopia grade > 0 and a reduction of ≥ 1 grade between baseline and the last infusion, and complete diplopia response defined as having baseline binocular diplopia grade > 0 and achieving grade of 0 as of the last infusion.
Quality of Life (QoL) as Reported by Participants | From baseline up to approximately 3 years
  All available participant-reported QoL for each participant, overall and at subscale level, and the change in QoL between baseline and the last infusion, overall and at subscale level.
Incidence of Adverse Events (AEs) | From baseline up to approximately 3 years
  The incidence of AEs between the administration of the first dose and 30 days after the last dose of teprotumumab, including:
  * Any AE
  * Specific AEs, inclusive of infusion-related reactions, hyperglycemia, hearing impairment, and new onset or exacerbation of IBD
  * Serious adverse event (SAE)
  * AE leading to treatment discontinuation
  * AE leading to death.
Status of Specific AEs up to 6 Months After Last Infusion of Teprotumumab | From baseline up to approximately 3 years
  Specific AEs include infusion-related reactions, hyperglycemia, hearing impairment, and new onset or exacerbation of IBD.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Boao Vanguard Hospital, Qionghai, Hainan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe, or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com